CLINICAL TRIAL: NCT05301881
Title: COntinue the SaMe Systemic Therapy After Local Ablative Therapy for Oligo Progression in Metastatic Breast Cancer - the COSMO Study
Acronym: COSMO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Maarten van de Weijden Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M21CSM
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer Invasive; Metastatic Cancer; Oligoprogressive
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Surgical Procedures, Operative; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Lesion(s) will be treated with surgery, radiotherapy or radiofrequent ablation depending on the location. The treatment is standard of care and will be decided in the treating team of the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Surgery, radiotherapy or radiofrequent ablation (Other): The oligoprogresive lesion(s) will be treated with Surgery, radiotherapy or radiofrequent ablation depending on the location of the lesion. treatment will be standard of care and will be decided by the treating team of the patient.
  Interventions: Procedure: Surgery; Radiation: Radiotherapy; Other: Radiofrequent ablation

INTERVENTIONS:
Procedure: Surgery — resection of the oligometastatic lesion(s)
Radiation: Radiotherapy — radiation of the oligometastatic lesion(s)
Other: Radiofrequent ablation — radiofrequent ablation of the oligometastatic lesion(s)

SUMMARY:
Patients with oligoprogression of metastatic breast cancer during palliative treatment that is amenable to local therapy will be included. The local ablative therapy (LAT) may consist of stereotactic ablative radiotherapy (SABR), also known as stereotactic body radiation therapy, surgery or radiofrequency ablation (RFA).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive breast cancer
* Metastatic breast cancer
* Oligoprogression defined as one or two distant metastatic lesions, limited to one organ, or the primary tumor or locoregional lymph nodes, increasing ≥20% in size and be larger than 15 mm or if metabolic activity increases (with 20% in SUVmax) on FDG-PET-CT.
* Systemic treatment can be either endocrine, targeted, chemotherapy or immune-checkpoint blockade
* Patients should be on systemic therapy for at least six months. Status should be stable disease or partial or complete response for at least 6 months.
* Oligoprogression has to be detected with radiological imaging comparing the lesion on the same type of imaging modality as has been used at the start of systemic therapy.
* The radiological imaging that shows progression must be performed within 70days prior to LAT.
* Bone metastases are classified as progressive if the lytic component of the lesion increases by ≥20% or the FDG-uptake increases by ≥20% on FDG-PET-CT
* Oligo-progression has to be confirmed with a FDG-PET-CT-scan 5-7 weeks after the initial scan that showed oligoprogression.
* Lesion(s) must be amenable to resection, radiotherapy or radiofrequency ablation with the intent of local obliteration
* Age ≥18
* World Health Organization (WHO) Performance Status 0 or 1
* Signed written informed consent before patient registration according to ICH/GCP, and national/local regulations

Exclusion Criteria:

* Having received more than two lines of systemic therapy for MBC If a treatment regimen has been de-escalated without adding other therapies, this is seen as one line of therapy. For example: Pertuzumab/trastuzumab+docetaxel followed by pertuzumab/trastuzumab will be viewed as one line of systemic therapy.
* Other malignancy except carcinoma in situ and basal-cell and squamous cell carcinoma of the skin, unless the other malignancy was treated ≥5 years ago with curative intent without the use of chemotherapy or radiation therapy
* Current pregnancy or breastfeeding. Women of childbearing potential must use adequate contraceptive protection
* Presence of any medical condition that would place the patient at unusual risk, up to the discretion of the clinician
* Presence of any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2035-04-01 (Estimated); Study Completion 2040-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients free of progression at 6 months | At 6 months
  progression-free survival at 6 months (PFS-6)

SECONDARY OUTCOMES:
Number of patients free of progression at 6 months per histoligical subtype | At 6 months
  PFS-6 for breast cancer subtypes: ER+/HER2- vs. HER2+ vs. TN
Number of patients free of progression at 6 months per breast cancer subtype | At 6 months
  PFS-6, stratified by breast cancer subtype
  - localization of progressive lesion
Number of patients free of progression at 6 months per localization of progressive lesion | At 6 months
  PFS at 6 months separately for localization of progressive lesion: locoregional vs. cranial vs. visceral vs. bone
Overall Surival (OS) | Up to 120 months
  Evaluation of overall survival measured from baseline till death due to any cause
Time to next line of treatment | Up to 120 months
  Time to next line of systemic therapy meeasured from baseline
Number of patients who develop "visceral crisis" | Up to 120 months
  number of patients who develop "visceral crisis"
Number of patients who develop complications after local ablative treatment | Up to 120 months
  Assess the number of patients who develop complications after local ablative treatment

CONTACTS AND LOCATIONS:
Overall Officials: G Sonke, Principal Investigator — The Netherlands Cancer Institute
Locations (7):
- Netherlands (7):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Antoni van Leeuwenhoek, Amsterdam
  - Rijnstate, Arnhem
  - Deventer ziekenhuis, Deventer
  - ADRZ, Goes
  - Martini ziekenhuis, Groningen
  - Antonius ziekenhuis, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided
to be determined